CLINICAL TRIAL: NCT00459056
Title: The Vascular Effects of Carvedilol Controlle Release (CR) + Lisinopril Versus Lisinopril + Hydrochlorothiazide (HCTZ) in Abdominally Obese Hypertensive Patients
Brief Title: The Vascular Effects of Carvedilol Controlled Release (CR) in Abdominally Obese Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Paul Heart Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Aaron S. Kelly, Ph.D., Assistant Professor, University of Minnesota
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPHC 2007-01
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-11

CONDITIONS: Abdominal Obesity; Hypertension
MeSH Terms: conditions — Obesity, Abdominal; Hypertension | interventions — Carvedilol; Lisinopril; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvediolol CR + Lisinopril, then Lisinopril + HCTZ (Experimental): Subjects were randomly assigned to Carvedilol CR + Lisinopril for three months, then had a washout period of one month, and then were given Lisinopril + HCTZ for the final three months.
  Interventions: Drug: Carvedilol CR + Lisinopril; Drug: Lisinopril + HCTZ
- Lisinopril + HCTZ, then Carvedilol CR + Lisinopril (Active Comparator): Subjects were randomally assigned to Lisinopril + HCTZ for three months, then had a washout period for one month, and then were given Carvedilol CR + Lisinopril for the final three months.
  Interventions: Drug: Carvedilol CR + Lisinopril; Drug: Lisinopril + HCTZ

INTERVENTIONS:
Drug: Carvedilol CR + Lisinopril — Participants were given Carvedilol CR + Lisinopril for three months. Oral medication. Carvedilol CR and Lisinopril combination therapy was initiated at 20 mg and 10 mg, respectively. Patients returned one week later and doses of carvedilol CR and lisinopril were increased to 40 mg and 20 mg, respectively, depending on blood pressure.
  Other Names: Prinivil; Coreg
Drug: Lisinopril + HCTZ — Participants were given Lisinopril + HCTZ for three months. Oral medication. Lisinopril + HCTZ combination therapy was initiated at 12.5 mg and 10 mg, respectively. Patients returned 1 week later and doses of hydrochlorothiazide and lisinopril were increased to 25 mg and 20 mg, respectively, depending on blood pressure levels.
  Other Names: Prinivil; Hydrochlorothiazide

SUMMARY:
The purpose of this study is to compare the effects of two different combination therapies for high blood pressure on vascular health.

DETAILED DESCRIPTION:
Hydrochlorothiazide (HCTZ) has been a popular choice for the treatment of hypertension mainly due to its efficacy in lowering blood pressure, safety, and cost-effectiveness. Similarly, angiotensin converting enzyme inhibitors (ACE-I), because of their neutral to positive impact on glycemic control, have been a popular choice for addressing hypertension in abdominally obese patients. Furthermore, the ACE-I drug class has been shown to improve vascular endothelial function and inflammation in addition to its blood pressure lowering effects.

Conversely, beta-adrenergic receptor blockers (b-blockers) have generally been avoided as first line anti-hypertensive therapy in pre-diabetic patients due to concerns about worsening glycemic control and potential hastening of progression to type 2 diabetes mellitus (T2DM). However, recent data have shown that the 3rd generation b-blocker carvedilol does not negatively affect glucose metabolism and therefore may be a safe and effective choice for blood pressure control in these patients. This neutral glycemic effect is likely due to the fact that carvedilol is a non-selective b-receptor antagonist (blocks both b1 and b2 receptors) with alpha1-receptor blocking properties. In addition, carvedilol possesses anti-oxidant properties and improves endothelial function, potentially making it an attractive anti-hypertensive treatment strategy in patients with abdominal obesity.

The combination of carvedilol and lisinopril may be especially effective in reducing blood pressure and may act synergistically to address the impaired vascular function and increased inflammation and oxidative stress present in patients with the metabolic syndrome phenotype. Therefore the primary objective of the current study will be to evaluate the effects of carvedilol CR + lisinopril compared to lisinopril + HCTZ on vascular function in a head to head trial in abdominally obese, hypertensive patients. The secondary objective will be to compare the effects of these two anti-hypertensive therapies on plasma biomarkers of endothelial activation, inflammation, and oxidative stress in these patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Systolic blood pressure (SBP) >130 and/or diastolic blood pressure (DBP) >85 (or currently taking anti-hypertensive medication)
* Waist circumference >102 cm (men) and >88 cm (women)
* Stable cardiovascular medication regimen (or other medications known to affect endothelial function) at least 1 month prior to enrollment and throughout the study

Exclusion Criteria:

* Use of anti-hypertensive medications within one month of randomization (patients may be washed-out from anti-hypertensive medications)
* Unstable angina
* History of angina symptoms within 3 months of screening
* Decompensated heart failure
* History of myocardial infarction
* Stroke or coronary artery bypass graft within 3 months of screening
* Standard clinical contraindications to beta-blocker therapy
* Standard clinical contraindications to ACE-I therapy
* Women who are currently pregnant or planning to become pregnant (pregnancy testing will occur at specific intervals throughout study and women will be informed of potential risks during the consenting process; information specific to this risk will be detailed in the consent form)
* Breastfeeding women
* Clinically significant liver disease
* Creatinine > 2.5 mg/dL
* Hepatic function greater than 3 times upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Kelly, PhD, Principal Investigator — St. Paul Heart Clinic
Locations (1):
- St. Paul Heart Clinic, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were recruited from medical clinics
Pre-assignment Details: Patients using anti-hypertensive medication(s) at baseline were allowed to undergo a 1-month washout prior to randomization.
Groups:
- Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ: Participants were randomized to Carvedilol CR + Lisinopril for three months, then had a one month wash-out period, and then were randomized to Lisinopril + HCT for the remaining three months. Carvedilol CR was initiated at a dose of 20mg, once per day, then titrated to 40mg, once per day after one week. Lisinopril was initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day after one week. For the second phase, lisinopril was again initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day, after one week. HCT was initiated at a dose of 12.5mg, once per day, then titrated to 25mg, once per day, after one week.
- Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril: Participants were randomized to Lisinopril + HCT for three months, then had a one month wash-out period, and then were randomized to Carvedilol CR + Lisinopril for the remaining three months. Lisinopril was initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day after one week. HCT was initiated at a dose of 12.5mg, once per day, then titrated to 25mg, once per day, after one week. For the second phase, Lisinophil was again initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day after one week. Carvedilol CR was initiated at a dose of 20mg, once per day, then titrated to 40mg, once per day after one week.
Period: First Intervention (First Three Months)
Arm/Group | Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ | Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril
Started | 10 | 15
Completed | 9 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Washout (1 Month)
Arm/Group | Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ | Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril
Started | 9 | 14
Completed | 9 | 14
Not Completed | 0 | 0
Period: Second Intervention (Final Three Months)
Arm/Group | Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ | Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril
Started | 9 | 14
Completed | 9 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ: Participants were randomized to Carvedilol CR + Lisinopril for the first three months, then had a washout period for one month, and then were given Lisinopril + HCTZ for the final three months.
- Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril: Participants were randomized to Lisinopril + HCTZ for the first three months, then had a washout period for one month, and then were given Carvedilol CR + Lisinopril for the final three months.
- Total: Total of all reporting groups
Arm/Group | Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ | Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril | Total
Number analyzed (Participants) | 10 | 15 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 25
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.21) | 54.9 (6.39) | 54.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Reactive Hyperemic Index by Period (Carvedilol CR + Lisinopril vs. Lisinopril + HCTZ)
Description: Reactive hyperemic index is a measure of endothelial function. This is measured by the ratio of post-occlusion blood volume flow versus the baseline blood volume flow. The outcome reported is the change in this ratio after the first intervention phase compared to after the second intervention phase.
Time Frame: Change from three months to seven months
Population: All completers were included in the analysis
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Carvedilol CR + Lisinopril, Then Lisinopril +HCTZ: Participants were randomized to Carvedilol CR + Lisinopril for the first three months, then had a one month washout period, then were given Lisinopril + HCTZ for the final three months. Carvedilol CR was initiated at a dose of 20mg, once per day, then titrated to 40mg, once per day after one week. Lisinopril was initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day after one week. For the second phase, lisinopril was again initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day, after one week. HCT was initiated at a dose of 12.5mg, once per day, then titrated to 25mg, once per day, after one week.
- Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril: Participants were randomized to Lisionopril +HCTZ for the first three months, then had a one month washout period, then were given Carvedilol CR + Lisinopril for the final three months. Lisinopril was initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day after one week. HCT was initiated at a dose of 12.5mg, once per day, then titrated to 25mg, once per day, after one week. For the second phase, lisinopril was again initiated at a dose of 10mg, once per day, then titrated to 20mg, once per day, after one week. Carvedilol CR was initiated at a dose of 20mg, once per day, then titrated to 40mg, once per day after one week.
Arm/Group | Carvedilol CR + Lisinopril, Then Lisinopril +HCTZ | Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril
Number analyzed (Participants) | 9 | 14
Ratio | -0.26 (0.59) | -0.14 (0.18)

ADVERSE EVENTS:
Time Frame: 7-months
Arm/Group | Carvedilol CR + Lisinopril, Then Lisinopril + HCTZ | Lisinopril + HCTZ, Then Carvedilol CR + Lisinopril
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/15
Other Adverse Events (participants affected / at risk) | 0/10 | 0/15

LIMITATIONS AND CAVEATS:
crossover study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No